CLINICAL TRIAL: NCT02939456
Title: Comparison Of Double Inversion Recovery Magnetic Resonance Imaging (Dir-Mri) And Dynamic Contrast Enhanced Magnetic Imaging (Dce-Mri) In Detection Of Prostate Cancer: A Pilot Study
Brief Title: Comparison Of DIR-MRI And DCE-MRI In Detection Of Prostate Cancer: A Pilot Study
Acronym: DIRMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1139
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2018-05

CONDITIONS: Cancer of the Prostate
Keywords: prostate; cancer; MRI
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DIR-MRI (Other): Participants will have Double Inversion Recovery Magnetic Resonance Imaging (DIR-MRI) as well as the standard Dynamic Contrast Enhanced Magnetic Imaging (DCE-MRI)
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Double Inversion Recovery Magnetic Resonance Imaging (DIR-MRI) and Dynamic Contrast Enhanced Magnetic Imaging (DCE-MRI)

SUMMARY:
This is a pilot study taking place at University Hospitals of North Midlands NHS Trust. Patients referred for MRI for possible prostate cancer will be invited to take part in the study. Following consent, participants will have an additional MRI sequence performed during their routine MRI called Double Inversion Magnetic Resonance Imaging (DIR-MRI).

Participants scan images and prostate biopsy histology report (if applicable) will be reviewed by the research team.

DETAILED DESCRIPTION:
This is a pilot study taking place at University Hospitals of North Midlands NHS Trust. Patients referred for MRI for possible prostate cancer will be invited to take part in the study. Following consent, participants will have an additional MRI sequence performed during their routine MRI called Double Inversion Magnetic Resonance Imaging (DIR-MRI). Participants scan images and prostate biopsy histology report (if applicable) will be reviewed by the research team. The research team will look at the variability of LNR score amongst the two scan typed and the DCE-MRI and DIR-MRI images will be correlated with biopsy results to give an indication of the accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for prostate MRI for possible prostate cancer
* Safe to undergo an MRI scan
* Able to give informed consent

Exclusion Criteria:

* MRI referrals where prostate cancer is not the question
* Patients who are not safe to undergo an MRI scan
* Patients who have undergone prostate biopsy in the previous 10 weeks
* Patients unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Lesion to Normal tissue Ratio (LNR) recorded for DIR-MRI and DCE-MRI | 3 months
  In order to inform a sample size calculation for a subsequent, fully powered equivalence trial Is DIR-MRI equivalent to DCE-MRI in detection of prostate cancer

SECONDARY OUTCOMES:
Correlation of biopsy and DIR-MRI and DCE-MRI findings | 3 months
  In order to ascertain if addition of DIR-MRI could improve accuracy of cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Onwuharine, Principal Investigator — University Hospitals of North Midlands NHS Trust
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No